CLINICAL TRIAL: NCT01214447
Title: Validity and Reproducibility of OSND (Objective Score of Nutrition on Dialysis) as a Nutritional Marker in End-stage Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Ilia Beberashvili MD, Nephrology Division, Assaf Harofeh Medical Center
Other Study IDs: 132/10
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Malnutrition-Inflammation Syndrome; Hemodialysis Nutritional Risk Stratification
Keywords: Hemodialysis; Inflammation; Malnutrition; Phase Angle
MeSH Terms: conditions — Inflammation; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Low - OSND less than 22
  Interventions: Other: No intervention
- Moderate - OSND score 23-27
  Interventions: Other: No intervention
- Normal - OSND score 28-32
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study - no intervention

SUMMARY:
This prospective observational study is planned to validate OSND against the prospective morbidity and mortality in chronic hemodialysis patients and to examine the hypothesis that OSND risk stratification of chronic HD patients is useful in predicting outcomes and better than its component alone or in diverse combinations. The investigators specific aim is to validate OSND in chronic HD patients by comparing it with conventional measures of nutritional state, including blood tests, anthropometry, MIS, GNRI, bioelectric impedance analysis and several measures of clinical outcome including prospective mortality and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18 years, in chronic hemodialysis treatment at least 3 months
2. Stable and adequate hemodialysis treatment three months prior to participation in study as defined by Kt/V > 1.2 and/or hemodialysis performed 4 hours 3 times weekly
3. Patients with normal hydration status (edema-free), with no neuroid-muscular diseases
4. Informed consent obtained before any trial-related activities

Exclusion Criteria:

1. Patients with edema, pleural effusion or ascites at their initial assessment
2. Patients with active malignant disease or liver cirrhosis
3. Patients with neuroid-muscular diseases
4. Patients on chronic treatment with steroids on doses > 10 mg/day Prednisone (or equivalent)
5. Patients treated with immunosuppressive agents
6. Patients suffering from

   * Acute vasculitis
   * Severe systemic infections
   * Heart failure (NYHA class III-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 stable chronic hemodialysis patients receiving maintenance hemodialysis treatment in our dialysis unit (nephrology division, Assaf Harofeh Medical Center) and in 2 satellite hemodialysis units (Nephromor, Rishon Lezion and Afek, Ramla).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
All cause morbidity and mortality | during 2 years of observation
  * Associations of OSND with:
    * Morbidity: Days at hospital (over night stay). Measured from baseline to end of study
    * Morbidity: Number of sick days during the study period
    * Morbidity: Number of visits to health care professionals other than hospitals
    * Mortality: From baseline visit to end of study
  * Interobserver reproducibility of OSND.

SECONDARY OUTCOMES:
All cause morbidity and mortality | 2 years
  Associations of MIS, GNRI and phase angle with:
  * Morbidity: Days at hospital (over night stay). Measured from baseline to end of study
  * Morbidity: Number of sick days during the study period
  * Morbidity: Number of visits to health care professionals other than hospitals
  * Mortality: From baseline visit to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ilia Beberashvili, MD, Principal Investigator — Nephrology division Assaf Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Background] Beberashvili I, Azar A, Sinuani I, Yasur H, Feldman L, Averbukh Z, Weissgarten J. Objective Score of Nutrition on Dialysis (OSND) as an alternative for the malnutrition-inflammation score in assessment of nutritional risk of haemodialysis patients. Nephrol Dial Transplant. 2010 Aug;25(8):2662-71. doi: 10.1093/ndt/gfq031. Epub 2010 Feb 26. PMID 20190238